CLINICAL TRIAL: NCT04678739
Title: Efficacy and Safety of Remdesivir and Tociluzumab for the Management of Severe COVID-19: A Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M Abdur Rahim Medical College and Hospital (Other Government)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other); Cox's Bazar 250 Bed District Sadar Hospital (Unknown); Chattogram General Hospital (Other Government)
Responsible Party: Principal Investigator, Abu Taiub Mohammed Mohiuddin Chowdhury, Resident, First Affiliated Hospital Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M.A.R.M.C.D./2020/1985
Record Dates: First submitted 2020-12-19; First posted 2020-12-22 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Covid-19 ARDS
Keywords: COVID 19; Remdesivir; Ticilizumab; COVID-19 ARDS
MeSH Terms: conditions — COVID-19 | interventions — remdesivir; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Remdesivir + Tocilizumab treatment group (Experimental): Drug: Remdesivir Injectable solution Tocilizumab Injectable solution A loading dose of Remdesivir I/V 5mg/kg (less than 40kg) or 200mg (>40kg) on day 1, then 2.5mg/kg (less than 40kg) or 100mg (>40kg) daily following randomization.
  Tocilizumab I/V 8mg/Kg up to 800mg highest 12 hours apart.
  Interventions: Drug: Remdesivir; Drug: Tocilizumab
- Group B: Control group (No Intervention): Treatment as given without Remdesivir and Tocilizumab.

INTERVENTIONS:
Drug: Remdesivir — Remdesivir 100 IV Infusion as a lyophilized powder
  Arms: Group A: Remdesivir + Tocilizumab treatment group
Drug: Tocilizumab — Actemra IV Infusion
  Other Names: Actemra IV Infusion
  Arms: Group A: Remdesivir + Tocilizumab treatment group

SUMMARY:
This randomized clinical trial was designed and intended to evaluate the efficacy of Remdesivir and Tocilizumab as a treatment for severe Acute Respiratory Distress Syndrome (ARDS) caused by Coronavirus disease 2019 (COVID-19). Our aim is to find the best option for the treatment and management of ARDS in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

Severe COVID-19 patients require hospitalization under HDU/ICU. The SARS-CoV-2 infection will be confirmed by RT PCR / CT Chest in every case.

Exclusion Criteria:

* Participants with uncontrolled clinical status who were hospitalized from the before.
* Contraindication / possible drug interaction.
* Participants who have any severe and/or uncontrolled medical conditions like, Severe ischemic heart disease, epilepsy, malignancy, Pulmonary/renal/hepatic disease, AIDS, Pulmonary TB, pregnancy, Corpulmonale, and etc.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Time to Clinical Improvement (TTCI) | Following randomization 30 days.
  Time to Clinical Improvement (TTCI) Defined as Time from Randomization to National Early Warning Score 2 (NEWS2) Score of </= 2 Maintained for 24 Hours.

SECONDARY OUTCOMES:
Duration of ICU Stay | Following randomization 30 days.
  Duration of ICU Stay in Days
Mortality Rate | Following randomization 30 days.
  Mortality Rate on Days during hospitalization
Time to Recovery | Following randomization 30 days.
  Defined as Time from Randomization to the Time when a Non-ICU Hospital Ward or not Requiring Supplemental Oxygen, or Better is Observed
Hospital stay | Following randomization 30 days.
  Time from Randomization to Hospital Discharge or "Ready for Discharge" (as Evidenced by Normal Body Temperature and Respiratory Rate, and Stable Oxygen Saturation on Ambient Air or </= 4L Supplemental Oxygen)
Rate of daily Supplemental Oxygen Use | Following randomization 30 days.
  Rate of daily Supplemental Oxygen Use by the patient
Time to Clinical Failure | Following randomization 30 days.
  Time to Clinical Failure, Defined as the Time from Randomization to the First Occurrence of Death, Mechanical Ventilation or Withdrawal (whichever occurs first)

CONTACTS AND LOCATIONS:
Overall Officials: Abu Taiub Mohammed Mohiuddin Chowdhury, MBBS, MD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University; Akter Kamal, MD, PhD, Study Director — M Abdur Rahim Medical College Hospital
Locations (3):
- Bangladesh (3):
  - Chattogram General Hospital, Chittagong
  - Cox's Bazar 250 Bed District Sadar Hospital, Cox’s Bāzār
  - M. Abdur Rahim Medical College Hospital, Dinajpur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohiuddin Chowdhury ATM, Kamal A, Abbas KU, Talukder S, Karim MR, Ali MA, Nuruzzaman M, Li Y, He S. Efficacy and Outcome of Remdesivir and Tocilizumab Combination Against Dexamethasone for the Treatment of Severe COVID-19: A Randomized Controlled Trial. Front Pharmacol. 2022 Apr 5;13:690726. doi: 10.3389/fphar.2022.690726. eCollection 2022. PMID 35450050